CLINICAL TRIAL: NCT06408961
Title: Extracellular Vesicle Signaling in Obesity and Cardiometabolic Disease (EVOC)
Brief Title: EVOC - EVs in Obesity and Cardiometabolic Disease
Acronym: EVOC
Status: Recruiting | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Collaborators: American Heart Association (Other)
Responsible Party: Principal Investigator, Saumya Das, Principal Investigator, Massachusetts General Hospital
Other Study IDs: 2022P002665
Record Dates: First submitted 2024-05-07; First posted 2024-05-10 (Actual); Last update posted 2025-11-13 (Actual); Status verified 2025-11

CONDITIONS: Cardiovascular Diseases
Keywords: Extracellular Vesicles; Cardiometabolic Disease; Cardiovascular Risk; Type II Diabetes
MeSH Terms: conditions — Cardiovascular Diseases; Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The study will be collecting plasma, subcutaneous fat tissue and visceral fat tissue.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Bariatric Surgery: Patients undergoing bariatric surgery

SUMMARY:
The goal of this observational study is to research the impact of molecular signals from the heart, liver and fat tissue on cardiovascular disease risk, and the presentation of Type II Diabetes and diseases that affect the heart, blood vessels and metabolism (Cardiometabolic Disease). Specifically, the focus is on the content and function of Extracellular Vesicles (EVs), small sacs released from a cell's surface that contain important molecular cargo. The main questions it aims to answer are:

1. What molecular cargo do adipose-tissue EVs carry?
2. How do these cargo impact cardiac and hepatic function?
3. Are changes in EV content related to cardiac function and adiposity with weight loss?

Tissue samples from fat tissue and blood samples will be collected from patients receiving bariatric weight loss surgery.

DETAILED DESCRIPTION:
The primary clinical objective of this research is to study the impact of molecular signals from the adipose tissue to the heart, liver and brain on cardiovascular disease risk in obesity, Type II Diabetes and other metabolic diseases that affect the heart, blood vessels and metabolism (Cardiometabolic Disease). Specifically, the focus is on the content and function of Extracellular Vesicles (EVs), small sacs released from a cell's surface that contain important molecular cargo. The hypothesis is that EVs derived from metabolically active fat tissue located around the abdominal organs (visceral adipose tissue) have a different cargo than those derived from non-metabolically active fat tissue located directly under the skin (subcutaneous adipose tissue), and that these cargoes impact the function of other organs. Further, we hypothesize that visceral adipose EVs are also present in the plasma in circulation, and that the content changes as patients become metabolically healthy following bariatric surgery.

After obtaining patient consent, samples from visceral fat tissue, subcutaneous fat tissue and blood will be collected during the gastric bypass weight loss surgery. These samples will be brought to lab where they will be processed for EVs. Subject's medical history and records will be followed as well. An optional, secondary blood draw may be collected 3 month post-surgery or within 24 months.

Following collection, the samples will be brough to the laboratory of the PI for processing. Samples will undergo characterization for proteins, extracellular or exosomal RNAs, tissue RNAs (e.g., leukocyte/buffy coat), and/or metabolites. A trascriptomic and proteomic analysis will be performed to determine differences in protein and RNA expression. The EVs will be extracted from subcutaneous and visceral fat tissue and used to treat heart muscle cells and liver-on-chip cells that have been produced in a laboratory setting.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 18 years of age
* Obese (BMI>/=30 kg/m2; for obesity/bariatric surgery group)
* For 20 patients, additional criteria will be presence of pre-diabetes or diabetes (HgbA1c > 5.7 or Fasting blood glucose > 100).

Exclusion Criteria:

* Pregnancy (as adjudicated by patient history)
* Prior clinical history of myocardial infarction or valvular heart disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of 100 eligible subjects with obesity (BMI>/=30 kg/m2) who are planned to undergo bariatric surgery recruited from the clinic of Dr. Denise Gee in the Weight Center at Massachusetts General Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-02-02 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
What are the contents inside of fat (adipose) tissue derived Extracellular Vesicles (EVs)? | 2 years
  The study staff aim to obtain EVs from fat samples obtained at the time of bariatric weight loss surgery. The activity of genes within the cargo of the collected EVs are assessed using RNA sequencing and protein contents analysis. A statistical analysis performed utilizing computer technology will provide us with differentially expressed cargo that may be a step in the molecular communication pathway to the heart and liver tissues.
How does the contents of Extracellular Vesicles (EVs) impact cardiac and liver function? | 2 years
  The study will look at the functional role of EVs from visceral and subcutaneous fat tissue on 3D organ on chip (liver on chip) and the heart's muscle cells (cardiomyocytes) using microscopes, gene expression and an assessment of the cardiomyocyte's electrical properties. It is predicted that changes in the recipient cell's gene expression will correlate with the contents discovered in Outcome 1.
Are changes in Extracellular Vesicle (EV) content related to cardiac function and adiposity with weight loss? | 2 years
  EVs collected from fat tissue are present in blood and provide a minimally invasive method to determine the fat cell's activity for turning food to into energy. We aim to assess how the content of EVs collected from plasma within the blood, and the content related to fat tissue EVs from Objective 1 change with weight loss.

SECONDARY OUTCOMES:
How does the presence of diabetes or pre-diabetes alter the RNA content of Extracellular Vesicles? | 2 years
  The fat samples will be categorized based on the presence of diabetes, pre-diabetes and no diabetes of the subject at the time of weight loss surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Saumya Das, MD, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Chatterjee E, Betti MJ, Sheng Q, Lin P, Emont MP, Li G, Amancherla K, Garcia-Contreras M, Gokulnath P, Limpitikul WB, Whittaker OR, Luong K, Azzam C, Gee D, Hutter M, Flanders K, Sahu P, Flynn CR, Brown J, Yu D, Rosen ED, Van-Keuren Jensen K, Gamazon ER, Shah R, Das S. The extracellular vesicle transcriptome provides tissue-specific functional genomic annotation relevant to disease susceptibility in obesity. Cell Genom. 2025 Sep 10;5(9):100925. doi: 10.1016/j.xgen.2025.100925. Epub 2025 Jul 15. PMID 40669467